CLINICAL TRIAL: NCT07253454
Title: Combined Use of Machine Learning and Metabolomics to Improve the Diagnosis and Management of Hyperandrogenism
Acronym: HYPERMETABO
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251139
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Hyperandrogenism
Keywords: fertility
MeSH Terms: conditions — Hyperandrogenism | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- principal group
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — collection of data from medical records over a period of 5 years

SUMMARY:
Hyperandrogenism is a common reason for consultation, the causes of which can range from common conditions (PCOS) to rarer conditions with major genetic implications (NC21OHD). It is characterized by elevated levels of circulating androgens, mainly testosterone. This excess of androgens usually manifests clinically as increased male-pattern hair growth and, less specifically, acne and alopecia. Its prevalence is estimated at between 6 and 12% in women of reproductive age, and its incidence is increasing.

It is also responsible for infertility. As a reminder, infertility is a major public health issue and affects more and more couples around the world.

The investigators therefore wish to develop innovative tools to improve the diagnosis and management of hyperandrogenism

DETAILED DESCRIPTION:
Hyperandrogenism is a common reason for consultation, the causes of which can range from common conditions (PCOS) to rarer conditions with major genetic implications (NC21OHD). It is characterized by elevated levels of circulating androgens, mainly testosterone. This excess of androgens usually manifests clinically as increased male-pattern hair growth and, less specifically, acne and alopecia. Its prevalence is estimated at between 6 and 12% in women of reproductive age, and its incidence is increasing.

It is also responsible for infertility. As a reminder, infertility is a major public health issue and affects more and more couples around the world.

The investigators therefore wish to develop innovative tools to improve the diagnosis and management of hyperandrogenism

ELIGIBILITY:
Inclusion Criteria:

* Patients of childbearing age (16 to 45 years old)
* Suffering from hyperandrogenism
* Established etiological diagnosis with elimination of differential diagnoses
* Informed and not opposed to the collection of their data for the purposes of the study

Exclusion Criteria:

* Pregnancy
* Patients under legal protection measures

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The first stage of the study will involve participating centers selecting patients' medical records after verifying their eligibility. It should be noted that the control group will consist of a population for whom tests were carried out for symptoms that were ultimately ruled out with normal results.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Use of machine learning models combined with metabolomics to distinguish between different causes of hyperandrogenism | 5 years

SECONDARY OUTCOMES:
Use of metabolomics to improve the management of patients with hyperandrogenism | 5 years
Use of metabolomics to predict CYP21A2 genotyping results | 5 years
Study of the impact of anti-androgenic hormone therapy on the predictive capabilities of the model | 5 years

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.